CLINICAL TRIAL: NCT00230256
Title: Treatment Outcomes and Quality of Life After IMRT Treatments of Head and Neck Cancers
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: ENT0003; ENT0003 (Other: Stanford University); 79057 (Other: Stanford University Secondary IRB Approval Number)
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the research study is to evaluate effectiveness and the quality of life, specifically the risk of dry mouth, after radiation treatment for head and neck cancers.

ELIGIBILITY:
Inclusion Criteria:Patients who complete radiation therapy for H&N cancers at Stanford University

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who complete radiation therapy for H&N cancers at Stanford University
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2003-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States